CLINICAL TRIAL: NCT02628197
Title: Effect of Periodontitis on Bone Mineral Density in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Perio 3 Aastha
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: PERIODONTITIS; Osteopenia
MeSH Terms: conditions — Periodontitis; Bone Diseases, Metabolic | interventions — Calcium; Vitamin D; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL GROUP (Active Comparator): 34 osteopenic postmenopausal women with chronic periodontitis who received calcium (500mg) and vitamin D (250I.U.) supplementation twice a day for 6 months.Scaling and root planing was not done in this group.
  Interventions: Dietary Supplement: calcium (500mg) and vitamin D (250I.U.)
- TEST GROUP (Active Comparator): 34 osteopenic postmenopausal women with chronic periodontitis who received scaling and root planing along with calcium (500mg) and vitamin D (250I.U.) supplementation twice a day for 6 months.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Dietary Supplement: calcium (500mg) and vitamin D (250I.U.) — calcium (500mg) and vitamin D (250I.U.) was given twice a day for 6 months
  Arms: CONTROL GROUP
Procedure: Scaling and root planing — scaling and root planing was done in the test group along with calcium (500mg) and vitamin D (250I.U.)
  Other Names: SRP
  Arms: TEST GROUP

SUMMARY:
The purpose of this interventional study was to investigate the impact of control of systemic inflammation by scaling and root planing (SRP) on bone mineral density (BMD) in osteopenic post-menopausal women with Chronic periodontitis(CP). Out of 68 osteopenic postmenopausal women with CP, 34 participants each were included in test and control group. BMD, hsCRP and periodontal parameters were recorded at baseline and 6 months.

DETAILED DESCRIPTION:
Rapid estrogen level decline after menopause is associated with systemic bone loss in women leading to osteopenia/osteoporosis. Estrogen therapy (ET) improves bone mineral density (BMD) in postmenopausal women. Currently, ET has been associated with statistically significant increased risk of breast cancer, stroke, and thromboembolic events. Easiest lifestyle modiﬁcation for the management of lower BMD is probably the adequate intake of calcium and vitamin D.

Chronic inflammatory diseases are associated with systemic bone loss. Bone has been a target in many inflammatory rheumatic diseases like rheumatoid arthritis (RA),and ankylosing spondylitis (AS). Low bone mineral density has also been documented in patients with Systemic lupus erythematosus (SLE).

Periodontitis is a chronic condition of supporting tissues of the teeth. It has been reported that 30% of individuals above the age of 50 years suffer from severe periodontitis.Hujoel et al has concluded that the mean periodontal surface area in patients with periodontitis can be as large as 8-20cm2 . The inflamed and ulcerated subgingival pocket epithelium may allow many gram negative and obligate anaerobic bacteria to enter bloodstream. Bacterial components such as endotoxins and major outer membrane proteins may also be disseminated. Studies on systemic influence of periodontitis have theorized that locally produced pro-inflammatory cytokines such as interleukin-1(IL-1), tumour necrosis factor-alpha(TNF-α), interleukin-6(IL-6) and prostaglandin-E2(PGE2) may be released into the circulation and exercise distant effects. These inflammatory cytokines have been reported to be implicated for the distinctive loss of bone density in osteoporosis through their effect on osteoclast activity.

C-reactive protein (CRP) is an extremely sensitive and non-specific acute phase reactant that is produced in response to tissue damage, inflammation, infection and hypoxia. It is a serological marker of systemic inﬂammation. Previous studies on elderly females and a large population based sample reported higher serum levels of CRP associated with lower BMD. A study also implicated that CRP ≥ 4.2mg/l may be used to identify the groups having rapid bone loss in older people. Various studies concluded higher levels of CRP in patients with periodontitis than in control. D Auito reported CRP reduction of 0.5mg/l at 6 months after non- surgical periodontal therapy in patients with chronic periodontitis(CP).Epidemiological studies from Buffalo, New York, reported elevated CRP in blood plasma among patients with severe periodontal attachment loss in comparison to individuals with minimal or no attachment loss. Various cross sectional studies have reported association between osteoporosis and periodontal disease in post-menopausal women. A recent study demonstrated that severe clinical attachment loss (CAL) was independently associated with low BMD of the femoral neck in postmenopausal women. These studies infer that osteoporosis is a risk factor for periodontitis. It is difficult to infer cause and effect relationship from cross sectional studies. The basis of association between osteoporosis and periodontitis may either be osteoporosis influencing periodontitis and/or vice-versa and/or both of them sharing common risk factors.

Inflammation has been reported to contribute towards post-menopausal deterioration in BMD. Levels of inflammatory cytokines responsible for the loss of bone density e.g. IL-1β, IL-6, TNF-α in osteoporosis are reported to be increased in the systemic circulation in CP. Hence, it is hypothesized that CP, an inflammatory disorder with a large wound surface area, may add to the systemic inflammatory burden and may consequently contribute towards deterioration of BMD in post-menopausal women. So, controlling systemic inflammatory burden by scaling and root planing(SRP) may have an adjunctive effect in the management of osteopenia/osteoporosis in these patients.

Taking into consideration these observations, the present study was undertaken to evaluate the impact of control of inflammation by SRP on BMD in osteopenic post-menopausal women with periodontitis.

MATERIALS AND METHODS Study Population Patients for this interventional study were recruited from the out-patient department of the department of Periodontics and Oral Implantology and department of Oral Medicine, Post Graduate Institute of Dental Sciences, Rohtak. The study protocol was carried out in accordance with the ethical standards outlined in the 1975 Declaration of Helsinki, as revised in 2013. The protocol was approved by the Institutional Review Board, Pt. B. D. Sharma University of Health Sciences, Rohtak and the ethical approval was obtained from the ethical committee of PGIDS, Rohtak. (PGIDS/IEC/2014/114). Prior written informed consent was taken from each patient after explaining the procedure along with the risks and benefits in their own language.

The patients accepted for the study met the following inclusion criteria: 1) osteopenic post-menopausal women with CP with 20 or more natural teeth (excluding third molars); 2) aged 52 -59 years; and 3) history of natural menopause since more than 5 years. Osteopenia criteria as per the World Health Organization (WHO) criteria : standardized T-score between -1.0 and -2.5 . CP criteria considered for the study were : at least 4 teeth on which one or more sites with a probing depth ≥ 4mm, CAL ≥ 3mm and the presence of bleeding on probing at the same site. Exclusion criteria included the following: 1) systemic disease known to affect BMD and hsCRP levels including RA, AS, SLE, IBD, COPD; 2) systemic disease known to affect the course of periodontal disease like diabetes mellitus or immunological disorder; 3) treatment with the following drugs in the previous 3 months: steroids, immune suppressants, antibiotics, anti-inflammatories, statins, lipid lowering drugs, anti-convulsants, thiazide diuretic agents, anti-coagulants or any other host modulatory drug; 4) recent history or presence of acute or chronic infection; 5) history of metabolic bone disease, thyroid and parathyroid disease and gastro-intestinal disorders; 6) early onset of menopause; treatment with systemic medication for osteoporosis/osteopenia including calcium and vitamin D supplementation, bisphosphonates etc.; 7) history of hysterectomy and hormone replacement therapy; 8) current or former smokers or use of smokeless tobacco in any form; and 9) periodontal treatment within past one year prior to inclusion into the study

STUDY GROUPS The test group consisted of 34 participants who received SRP along with calcium (500mg) and vitamin D (250I.U.) supplementation (Shelcal, torrents pharmaceutical limited, Gujarat, India) twice a day for 6 months while the control group consisted of 34 participants who received calcium (500mg) and vitamin D (250I.U.) supplementation* twice a day for 6 months. Participants without any chief complaint with reference to periodontitis who expressed their inability to undergo periodontal treatment immediately in near future were included in the control group.

BMD measurement BMD of the participants was evaluated using Dual Energy X-ray Absorptimetry( DXA, Hologic QDR explorer version 12.6:3; Hologic Inc., Bedford, MA, USA) in lumbar spine region (L1-L4) with an exposure of .07mGy for 90 seconds at baseline and 6 month follow-up. The improvement in BMD (T-score) at 6 months from baseline was taken as primary outcome.

Sample collection All the blood samples were collected at baseline and 6 month follow-up for serum high-sensitivity C - reactive protein (hsCRP). Venous blood from anticubital vein was collected after applying tourniquet in plain vacutainer tube without additive. It was measured using serum samples.

hsCRP estimation Serum hsCRP levels were assessed using a kit with high-sensitivity methodology‡( C - reactive protein (Latex) High-Sensitive Assay, Roche Diagnostics, GmbH, Mannheim, USA) in an autoanalyser according to manufacturer's instructions. The test principle was particle enhanced immune-turbidimetric assay, in which human CRP agglutinates with latex particles coated with monoclonal anti-CRP antibodies. The turbidity induced by the formation of immune complexes was measured at 546 nm.

Periodontal examination After their selection for the study, all participants underwent full-mouth periodontal examination at baseline and 6 month in a standardized way using illumination by a standard dental light, a mouth mirror, tweezer, manual calibrated probe( PCP-UNC 15 Hu-Friedy, Chicago, IL, USA) and explorer. Following parameters were taken into consideration: Plaque index (PI)(Silness & Loe); Gingival index (GI)(Loe & Silness); Bleeding on probing (BOP); Pocket depth (PD); and Attachment loss (AL). To preclude inter examiner variability, periodontal examination was performed by one trained and calibrated examiner (AB). The calibration protocol included determination of examiner reproducibility, which was recorded twice at the same visit on 10% of representative samples. Operator calibration for GI was based on intra examiner exact reproducibility at 85% of sites. For PD and AL, calibration was based on intra-examiner reproducibility within 1 mm at >90% and >85% of sites.

Periodontal treatment Patients in TG received full mouth scaling and root planing (SRP) using manual instruments and ultrasonic scaler (Suprasson P5 Booster; Satelec, Merignac Cedex, France) in 2-4 sessions. The patients were further provided information on the periodontal disease, and oral hygiene instructions were given at each appointment. The patients were instructed to use only mechanical techniques such as toothbrushes and interdental-floss during the study period. Mouthwashes and /or antimicrobials were not prescribed. Patients were asked to bring the remaining tablets left with them so as to assess the compliance. Patient compliance was considered when ≥90% of the tablets was consumed. Weekly reminders were also given to the patients through personal phone calls.

Statistical analysis Post-hoc analysis was done using statistical software (G*Power v.3.0.10, Heinrich-Heine University Düsseldorf, Düsseldorf, Germany). Effect size was determined following rule of the standardized difference in a given output variable (BMD) with sample size of 62 with significance level of two sided α= 0.05. This came out to be 1. With these measurements, statistical power exceeds 90% with allocation ratio of 1:1. The normality of the data distribution was examined using Shapiro-wilk test. PD and hsCRP were found to be normally distributed, whereas rests of the parameters were non-normally distributed. The descriptives were expressed as mean±SD. The significance of difference between groups for age, BMD, PI, GI, BOP and AL at baseline was compared by Mann-whitney U test. Independent T test was used in hsCRP and PD for the same purpose. Wilcoxon signed rank test and Paired T test were used to evaluate difference between baseline and 6 month follow up in both groups. The difference between groups was assessed using Mann whitney U test or Independent T test whichever was applicable. A binomial logistic regression model was fitted to relate Normal T-score patients as the outcome variable and treatment groups as the categorical predictor variable. The Hosmer-Lemeshow goodness of fit test was applied to verify whether the present test fits well. Model was adjusted for the covariate and all statistical analyses were 2 tailed, having a significance level at 0.05(SPSS v.21, IBM, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

1. osteopenic post-menopausal women with CP with 20 or more natural teeth (excluding third molars)
2. aged 52 -59 years
3. history of natural menopause since more than 5 years. Osteopenia criteria as per the World Health Organization (WHO) criteria : standardized T-score between -1.0 and -2.5 .

   * CP criteria considered for the study were : at least 4 teeth on which one or more sites with a probing depth ≥ 4mm, CAL ≥ 3mm and the presence of bleeding on probing at the same site.

Exclusion Criteria:

1. systemic disease known to affect BMD and hsCRP levels including RA, AS, SLE, IBD, COPD
2. systemic disease known to affect the course of periodontal disease like diabetes mellitus or immunological disorder
3. treatment with the following drugs in the previous 3 months: steroids, immune suppressants, antibiotics, anti-inflammatories, statins, lipid lowering drugs, anti-convulsants, thiazide diuretic agents, anti-coagulants or any other host modulatory drug
4. recent history or presence of acute or chronic infection
5. history of metabolic bone disease, thyroid and parathyroid disease and gastro-intestinal disorders
6. early onset of menopause; treatment with systemic medication for osteoporosis/osteopenia including calcium and vitamin D supplementation, bisphosphonates etc.
7. history of hysterectomy and hormone replacement therapy
8. current or former smokers or use of smokeless tobacco in any form
9. periodontal treatment within past one year prior to inclusion into the study

Ages: 52 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
bone mineral density | 6 months